CLINICAL TRIAL: NCT05482672
Title: GetHealthy-OA: A Biopsychosocial Treatment Approach to Improve Pain and Function for Patients With Comorbid Knee Osteoarthritis, Obesity, and Depression
Brief Title: GetHealthy-OA: A Program to Improve Pain and Function for Patients With Knee Osteoarthritis, Obesity, and Depression
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Cale Andrew Jacobs, PhD (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Cale Andrew Jacobs, PhD, Invetigator, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 80389
Record Dates: First submitted 2022-07-26; First posted 2022-08-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis; Obese; Depression
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity; Depression | interventions — fisetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study pharmacist that prepared the randomization schedule will meet with the pre-specified unblinded study personnel prior to the site initiation visit. The unblinded personnel will then prepare sealed envelopes that contain each subject's group assignment.
  The investigators will designate, a priori, study personnel that will be unblinded. These unblinded personnel will be directly involved with maintaining the drug log and communicating with participants to schedule virtual mind-body sessions. The unblinded pharmacist/coordinator will access the actual treatment assignment but both blinded study personnel and the patient will not know the patient's treatment assignment. The Investigator, participant, patient assessors, laboratory personnel, and statistician will remain blinded throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GetHealthy-OA (Experimental): The GetHealthy-OA program combines a 6-week mind-body program delivered via live video with the oral supplement fisetin. Oral fisetin will be taken for 2 consecutive days (day 1 and 2), a 28-day wash-out period, and then another 2-day course (days 31 and 32).
  Interventions: Drug: Fisetin; Behavioral: GetHealthy-OA mind-body program
- Minimally Enhanced Usual Care (Placebo Comparator): The minimally enhanced usual care group will be given a health education booklet at the date of baseline testing and will take an oral placebo for 2 consecutive days (day 1 and 2) and then again 28 days later (days 29 and 30).
  Interventions: Drug: Placebo oral capsule; Behavioral: Health education booklet

INTERVENTIONS:
Drug: Fisetin — Fisetin is a plant flavanol senolytic found in strawberries, persimmons, and cucumbers. This naturally derived senolytic has few side effects and previous animal models of both osteoarthritis and rheumatoid arthritis have demonstrated that the senolytic supplement fisetin reduces inflammation and slows cartilage breakdown.
  Other Names: Novusetin; 7,3',4'-flavon-3-ol; 3,3',4',7-tetrahydroxyflavone
  Arms: GetHealthy-OA
Behavioral: GetHealthy-OA mind-body program — The GetHealthy-OA mind-body program emphasizes increased physical activity, healthy diet and sleep habits to lessen osteoarthritis and depressive symptoms
  Arms: GetHealthy-OA
Drug: Placebo oral capsule — The oral placebo will consist of corn starch and gelatin capsules
  Arms: Minimally Enhanced Usual Care
Behavioral: Health education booklet — The booklet will containing brief summarized information that reflects the active intervention topics including the trajectory of pain and recovery for those with knee osteoarthritis, the role of relaxation strategies to manage pain, and the importance of returning to engagement in activities of daily living
  Arms: Minimally Enhanced Usual Care

SUMMARY:
The investigators have previously identified knee osteoarthritis patients with the combination of depression and an unhealthy weight may be an increased risk of more rapid joint degeneration and worsening pain. The GetHealthy-OA program combines a mind-body program with the oral supplement fisetin to potentially reduce the risk for this population by treating psychosocial, mechanical, and inflammatory mechanisms of knee osteoarthritis. This randomized clinical trial will compare the GetHealthy-OA program to minimally-enhanced usual care plus an oral placebo.

DETAILED DESCRIPTION:
The study will employ a double-blind, randomized, placebo-controlled clinical trial to compare the the multimodal GetHealthy-OA program versus placebo. As part of this clinical trial, 120 patients will be randomized to 1 of 2 groups: The GetHealthy-OA program that combines a mind-body program with oral fisetin versus a control group treated with an oral placebo and minimally-enhanced usual care (MEUC). The GetHealthy-OA group will participate in the 6-week the mind-body program and will take oral fisetin for 2 consecutive days (day 1 and 2), a 28-day wash-out period, and then another 2-day course (days 31 and 32). The MEUC group will be given a health education handout at the date of baseline testing and will take an oral placebo for 2 consecutive days (day 1 and 2) and then again 28 days later (days 29 and 30). To determine if immediate improvements are realized and whether gains are sustained after the completing the program, participants will be assessed at baseline, 6 weeks, 3 months, and 6 months.

The GetHealthy-OA mind-body program is a live-video, group program delivered via secure telehealth with mind-body skills to reduce pain and increase physical activity to promote optimal joint loading. The on-line program will be delivered remotely by a psychologist based at Massachusetts General Hospital via Zoom and we will assess symptoms and monitor any technical difficulties. The program consist of 6 sessions that will last about 45 minutes. The sessions are done on your smartphone or computer, and will include a group of 4 to 5 other people with knee arthritis who are also taking part in the study with you at the same time. The GetHealthy-OA group will participate in the 6-week the mind-body program and will take oral fisetin for 2 consecutive days (day 1 and 2), a 28-day wash-out period, and then another 2-day course (days 31 and 32).

The MEUC group will be given a health education booklet at the date of baseline testing and will take an oral placebo (corn starch) for 2 consecutive days (day 1 and 2) and then again 28 days later (days 29 and 30). The booklet will contain brief summarized information that reflects the active intervention topics including the trajectory of pain and recovery for those with knee osteoarthritis, the role of relaxation strategies to manage pain, and the importance of returning to engagement in activities of daily living. The MEUC will be given an oral placebo (corn starch) that is identical to the fisetin capsules with the same dosing regimen as the GetHealthy-OA group. Similar to participants in GetHealthy-OA group, participants in this group will receive usual medical care as determined by the medical team. Usual care involves meetings with physicians, medical staff, and physical therapy. Usual care is identical in intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate knee osteoarthritis (Kellgren/Lawrence Grade II or III)
* Obesity (Body Mass Index > 30 kg/m2)
* History of concurrent psychotropics for < 2 weeks prior to initiation of treatment or on stable doses for > 6 weeks
* Access to an internet-enabled computer/smart phone
* Willingness to comply with the study protocol and assessments
* Cleared by a medical doctor to participate

Exclusion Criteria:

* Rheumatoid arthritis
* History of cancer within 5 years of screening; unable to walk/wheelchair-bound
* Prior surgical fixation of a femur or tibia fracture
* Taking high doses of opioid pain medication (>50 milligrams of morphine equivalent per day)
* Diagnosis of a medical illness expected to worsen in the next 6 months (e.g., malignancy)
* Active suicidal ideation or past-year psychiatric hospitalization; non-English speaking
* Lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder
* Current substance abuse or dependence (or a history within the past 6 months)
* Practice of yoga/meditation, or other mind body techniques once per week > 45 min within the last 3 months
* Engagement in regular moderate or vigorous physical exercise for >30 min daily
* Reduced or altered capacity due to administration of any mind-altering substances such as tranquilizers, conscious sedation or anesthesia, or brain injury
* Females who are nursing, pregnant or planning to become pregnant during the duration of study drug dosing
* Females or males who do not wish to abstain from sex or use contraceptive protection during study drug dosing and for 2 weeks after the last dose

  o Those not willing to use 2 of the following effective forms of contraception: sterilization surgery, intrauterine device (IUD), implantable rod, contraceptive shot/injection, oral contraceptives, patch, vaginal ring, diaphragm with spermicide, sponge with spermicide, cervical cap with spermicide, and/or a male or female condom
* Subjects who do not have the capacity to consent themselves
* Subjects who are unable to tolerate oral medication
* Subjects having previously undergone any of the following treatments in the stated time window.

  * Surgery on the Study Knee in the past 6 months
  * Partial or complete joint replacement in the study knee. Partial or complete joint replacement in the contralateral knee is acceptable as long as the surgery was performed at least 6 months prior to enrollment and the operative knee is asymptomatic
  * Patients who have undergone arthroscopic surgery (including microfracture and meniscectomy) on the Study Knee in the last 2 years prior to the Screening visit or are anticipated to have arthroscopic surgery on either knee at any time during the study period
  * Currently taking Losartan
  * Currently taking Warfarin or related anticoagulants
  * Senolytic agents taken within the past 6 months and are not willing to discontinue these medications through the duration of the study, including: Fisetin, Quercetin, Luteolin, Dasatinib, Piperlongumine, or Navitoclax
  * Drugs that induce significant cellular stress and are not willing to discontinue these medications through the duration of the study, including alkylating agents, anthracyclines, platins, other chemotherapy drugs
  * Medications that are sensitive substrates or substrates with a narrow therapeutic range for cytochrome P450 family 1 subfamily A member 2 (CYP1A2), cytochrome P450 family 2 subfamily C member 8 (CYP2C8), cytochrome P450 family 2 subfamily C member 9 (CYP2C9), cytochrome P450 family 2 subfamily C member 19 (CYP2C19), cytochrome P450 family 2 subfamily D member 6 (CYP2D6), cytochrome P450 family 3 subfamily A member 4 (CYP3A4), Organic Anion Transporting Polypeptide 1B1 (OATP1B1) or strong inhibitors or inducers of Cytochrome P450 3A4 (CYP3A4; e.g. cyclosporine, tacrolimus or sirolimus)
  * Subjects taking the following other drugs if they cannot be held (per the Medical Director Austin Stone, MD, PhD) for at least 2 days before and during administration of Fisetin: cyclosporine, tacrolimus, repaglinide, and bosentan
  * Significant liver disease (i.e. greater than or equal to 2x the upper limit of normal bilirubin levels) or as in the opinion of the Medical Director
  * Significant renal disease (estimated glomerular filtration rate (eGFR) of <60 ml/min/1.73m2) or as in the opinion of the Medical Director
  * History of other formally diagnosed joint diseases including osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Cushing's syndrome, Stickler's syndrome, joint infection, hemophilia, hemochromatosis, or neuropathic arthropathy of any cause
  * Patients with type 1 or 2 diabetes (Hemoglobin A1c (HbA1c) > 6.5%) and/or taking medications that affect insulin levels, including: Metformin (within the last week), Glucocorticoids (within the last month), Acarbose (within the last week)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario and MacMaster Universities Osteoarthritis Index (WOMAC) | Change between Baseline and 3 months
  The WOMAC is a self-administered questionnaire consisting of 24 items that is widely used in the evaluation of Hip and Knee Osteoarthritis. Scores range from 0 to 96 with lower scores being indicative of less severe osteoarthritis symptoms
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference | Change between Baseline and 3 months
  The PROMIS Pain Interference (Short Form 8a v1.0) assesses the consequences of pain on relevant aspects of a person's life including the extent to which pain limits engagement with social, cognitive, emotional, physical, and recreational activities. Scores range from 0 to 100 with greater scores indicative of greater pain interference
Change in Average Daily Step Count | Change between Baseline and 3 months
  ActiGraph wGT3X-BTLink accelerometer (ActiGraph, LLC, Fort Walton Beach, FL, USA) will be used to assess average step count over a 7-day period at baseline and the 3 post-intervention time points. This accelerometer is widely used to ecologically assess physical functioning outcomes in chronic pain and older adult trials

SECONDARY OUTCOMES:
Change in serum Interleukin-17 (IL-17) | Change between Baseline and 6-weeks, 3-months, and 6-months
  IL-17 has been associated with cellular senescence in osteoarthritis, with greater concentrations associated with increased senescent cell activity
Change in serum IL-4 | Change between Baseline and 6-weeks, 3-months, and 6-months
  IL-4 has been associated with cellular senescence in osteoarthritis, with reduced concentrations associated with increased senescent cell activity
Change in urinary C-terminal crosslinked telopeptide type II collagen (CTX-II) | Change between Baseline and 6-weeks, 3-months, and 6-months
  Urinary CTX-II has been identified as a biomarker for the diagnosis, staging, and evaluating the prognosis of hip and knee osteoarthritis
Change in serum Chondroitin Sulfate epitope 846 (CS846) | Change between Baseline and 6-weeks, 3-months, and 6-months
  CS846 is a marker of aggrecan synthesis and is elevated in the serum for those with osteoarthritis.
Change in Pain Numerical Rating Scale | Change between Baseline and 6-weeks, 3-months, and 6-months
  Consistent with other osteoarthritis trials, patients will be asked to report their average pain over the past 24 hours. Scores range from 0 (no pain) to 10 (extreme pain)
Change in Walking Speed | Change between Baseline and 6-weeks, 3-months, and 6-months
  The 40 m walk test will be used to assess walking speed and is recommended by OARSI for the assessment of OA. Increased times are associated with slower walking speed
Arthritis Self-Efficacy Scale (ASES) | Change between Baseline and 6-weeks, 3-months, and 6-months
  The ASES assesses arthritis-specific self-efficacy on a 20-item scale. The ASES contains pain (5 items), function (9 items) and other symptoms (6 items) that are scored on a very uncertain (1) to very certain (10) scale. Scores are calculated for 3 subscales (pain, function, other) and range from 1 to 10 and higher average scores indicate greater arthritis-specific self-efficacy
PROMIS Depression | Change between Baseline and 6-weeks, 3-months, and 6-months
  The PROMIS Depression (Short Form v1.08b) assesses depressive symptoms. Scores range from 0 to 100 with greater scores indicative of worse depressive symptoms
PROMIS Anxiety | Change between Baseline and 6-weeks, 3-months, and 6-months
  The PROMIS Anxiety (Short Form v1.08a) assesses symptoms of anxiety. Scores range from 0 to 100 with greater scores indicative of worse symptoms of anxiety
Pain Catastrophizing Scale (PCS) | Change between Baseline and 6-weeks, 3-months, and 6-months
  The PCS assesses hopelessness, helplessness, and negative rumination about pain on a 13-item scale. Higher scores (range = 0 to 52) indicate greater pain catastrophizing
RU SATED | Change between Baseline and 6-weeks, 3-months, and 6-months
  Sleep health is a multidimensional construct, and sleep disturbance is closely tied with knee OA pain and depressive symptoms. We will quantify sleep health using the six-item RU-SATED which is a validated instrument to quantify sleep health, and has been used in populations of older adults. Score range from 0 to 12, with higher scores associated with better sleep health

CONTACTS AND LOCATIONS:
Overall Officials: Cale Jacobs, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - UK Healthcare at Turfland, Lexington, Kentucky
  - UK HealthCare Joint Reconstruction and Replacement, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No